CLINICAL TRIAL: NCT04356599
Title: Prediction and Unraveling of Delayed Cerebral Ischemia in Patients With Subarachnoid Hemorrhage Using Early Dynamic 18F-FDG PET/CT Assessment of Cerebral Glucose Uptake (PREDISP)
Brief Title: Prediction of Delayed Cerebral Ischemia After Subarachnoid Hemorrhage Using Dynamic 18F-FDG PET/CT
Acronym: PREDISP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL19_0408
Record Dates: First submitted 2020-04-15; First posted 2020-04-22 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Aneurysmal Subarachnoid Haemorrhage
Keywords: Aneurysmal subarachnoid haemorrhage; Delayed Cerebral Ischemia; Positron emission tomography; Cerebral microcirculation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): All participants will receive study intervention
  Interventions: Other: Early dynamic 18F-FDG PET/CT assessment of cerebral glucose uptake

INTERVENTIONS:
Other: Early dynamic 18F-FDG PET/CT assessment of cerebral glucose uptake — The intervention will consist in a dynamic cerebral 18F-FDG PET study performed at D2+/-1. Kinetic modeling will be performed using in-house software at the global, regional, and voxel level. In addition, cerebral perfusion and blood-brain-barrier permeability will be assessed at D4+/- 1 using perfusion MRI and permeability MRI.

SUMMARY:
A pilot trial for assessing early microvascular alterations after aneurysmal subarachnoid hemorrhage using dynamic 18F-FDG PET/CT. The primary endpoint will be the measure of early changes in cerebral glucose uptake reflecting microperfusion.

DETAILED DESCRIPTION:
We hypothesize that an early irreversible microvascular deterioration following initial bleeding could contribute to DCI occurrence. More precisely, we suspect that DCI areas are somehow overlaps of regions in which microperfusion is precociously altered, shortening circulatory reserves, and territories of secondarily spasmed arteries further lowering blood flow, resulting in ischemia. We aim to explore the potential microvasculature alteration through cerebral glucose perfusion and metabolism assessment using early dynamic 18F-fluorodesoxyglucose Positron Emission Tomography/Computer Tomography (dynamic 18F-FDG PET/CT). If our hypothesis turned out to be valid, we would at the same time be able to determine risk factors for this unpredictable complication and gain remarkable insight into DCI pathophysiology. Thus, the purpose of this trial is to demonstrate, in patients affected by SAH, the correlation between early cerebral glucose uptake defects in 18F-FDG PET/CT and delayed cerebral infarction in magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* written informed consent to participate in the study must be obtained from the subject or proxy/legal representative prior to enrollment.
* males and females aged 18 years and older.
* SAH proven by computed tomography (CT) and that has occurred within the last 72 hours.
* ruptured saccular aneurysm angiographically confirmed by digital subtraction angiogram or CT angiogram, which has been successfully secured by surgical clipping or endovascular coiling.
* high-risk subjects for DCI: "thick clot" on the hospital admission CT (grade 3 or grade 4 on the modified Fisher Scale).
* a woman of childbearing potential is eligible only if the serum pregnancy test performed during the screening period is negative.

Exclusion Criteria:

* PET/CT contradications
* MRI contradications
* gadolinium or meglumine hypersensitivity
* glomerular filtration rate <30mL/min
* SAH due to other causes than ruptured saccular aneurysm.
* post-HSA cardiac arrest.
* high sustained ICP ( >20mmHg lasting >20min) despite optimal treatment.
* significant and concomitant organ failure amongst the following: hypotension with systolic blood pressure <90mmHg refractory to treatment; unresolved pulmonary edema or pneumonia with severe hypoxia defined as PaO2/FiO2 <150; severe cardiac failure requiring inotropic support.
* patients with "do-not-resuscitate" orders, withdrawal of care situation, dying patient.
* vulnerable patient populations (minor, legal vulnerability, prisoner)
* pregnant and nursing mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Quantification of K1 parameter. | Day 2 +/- 1 day after the initial bleeding
  A kinetic modeling for cerebral glucose uptake will be performed using in-house software in order to provide the K1 parameter (in min-1) in every voxel reflecting the cerebral blood flow (in mL/min).
Quantification of Ki parameter. | Day 2 +/- 1 day after the initial bleeding
  A kinetic modeling for cerebral glucose uptake will be performed using in-house software in order to provide the Ki parameter (in min-1) in every voxel reflecting the cerebral metabolic rate of glucose in µmol/100g/min.

SECONDARY OUTCOMES:
Delayed cerebral ischemic regions. | From day 2 to day 21 +/- 3 days after the initial bleeding
  Delayed cerebral ischemic lesions will be ascertained by routine MRI scans until the end of the period of time in which the subject may present DCI (D21+/-3).
Delayed spasmed arteries territories. | From day 2 to day 21 +/- 3 days after the initial bleeding
  Occurence of vasospasm will be determined on routine angiograms until the end of the period of time in which the subject may present vasospasm (D21+/-3).
Quantification of cerebral blood flow using DSC-MRI | At day 4 +/- 1 day after the initial bleeding
  Cerebral blood flow in mL/100g/min will be measured using DSC-MRI (Dynamic Susceptibility Contrast Magnetic Resonance Imaging)
Quantification of cerebral blood flow using ASL-MRI | At day 4 +/- 1 day after the initial bleeding
  Cerebral blood flow in mL/100g/min will be measured using ASL-MRI (Arterial Spin Labelling Magnetic Resonance Imaging)
Quantification of blood-brain-barrier permeability using DSC-MRI | At day 4 +/- 1 day after the initial bleeding
  The blood-brain barrier permeability will be measured using DSC-MRI. A kinetic modeling will be performed in order to provide the leakage parameter K2 (in min-1) in every voxel.
Quantification of blood-brain-barrier permeability using DCE-MRI | At day 4 +/- 1 day after the initial bleeding
  The blood-brain barrier permeability will be measured using DCE-MRI (Dynamic Contrast-Enhanced Magnetic Resonance Imaging). A kinetic modeling will be performed in order to provide the leakage parameter Ktrans (in min-1) in every voxel.

CONTACTS AND LOCATIONS:
Overall Officials: Kévin CHALARD, M.D., Principal Investigator — UH Montpellier
Locations (1):
- Département d'Anesthésie-Réanimation Gui de Chauliac 80 Av Augustin.Fliche, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 12 months after the main publication
Access Criteria: Data are provided to qualified investigators free of charge. Required documents to request data include a summary of the research plan, request form, and IRB review. Dataset will be shared after careful examination by the study board of investigators.